CLINICAL TRIAL: NCT04600505
Title: A Randomized, Single Blind, 3-Period, 3-Treatment, Single-dose, Crossover Study to Assess the Relative Bioavailability of BGF Propellant 1 and BGF Propellant 2 Compared With BGF MDI HFA in Healthy Subjects
Brief Title: A Study to Assess Drug Absorption of Fixed Dose Combinations of Budesonide, Glycopyrronium, and Formoterol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: D5985C00001
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Results first posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2022-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Budesonide; Glycopyrronium; Formoterol; Hydrofluoroalkane; Metered dose inhaler
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Masking Description: This is a single blind study with regard to BGF MDI treatment, administered with 3 different propellants (Treatment A, B or C), in which the participants will remain blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment Sequence ABC (Experimental): Participants will be randomized to one of the 6 different treatment sequences. Each participant will receive 3 single-dose treatments of BGF MDI (Treatment A; Treatment B; Treatment C) in 3 treatment periods, with first dose on Day -1 for all treatment periods.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Treatment Sequence BCA (Experimental): Participants will be randomized to one of the 6 different treatment sequences. Each participant will receive 3 single-dose treatments of BGF MDI (Treatment B; Treatment C; Treatment A) in 3 treatment periods, with first dose on Day -1 for all treatment periods.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Treatment Sequence CAB (Experimental): Participants will be randomized to one of the 6 different treatment sequences. Each participant will receive 3 single-dose treatments of BGF MDI (Treatment C; Treatment A; Treatment B) in 3 treatment periods, with first dose on Day -1 for all treatment periods.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Treatment Sequence ACB (Experimental): Participants will be randomized to one of the 6 different treatment sequences. Each participant will receive 3 single-dose treatments of BGF MDI (Treatment A; Treatment C; Treatment B) in 3 treatment periods, with first dose on Day -1 for all treatment periods.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Treatment Sequence BAC (Experimental): Participants will be randomized to one of the 6 different treatment sequences. Each participant will receive 3 single-dose treatments of BGF MDI (Treatment B; Treatment A; Treatment C) in 3 treatment periods, with first dose on Day -1 for all treatment periods.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Treatment Sequence CBA (Experimental): Participants will be randomized to one of the 6 different treatment sequences. Each participant will receive 3 single-dose treatments of BGF MDI (Treatment C; Treatment B; Treatment A) in 3 treatment periods, with first dose on Day -1 for all treatment periods.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C

INTERVENTIONS:
Drug: Treatment A — Participants will receive 2 inhalations of BGF MDI with propellant 1.
  Other Names: BGF MDI Propellant 1
Drug: Treatment B — Participants will receive 2 inhalations of BGF MDI with propellant 2.
  Other Names: BGF MDI Propellant 2
Drug: Treatment C — Participants will receive 2 inhalations of BGF MDI with HFA propellant.
  Other Names: BGF MDI HFA

SUMMARY:
The study will evaluate bioavailability, pharmacokinetics, safety, and tolerability of budesonide, glycopyrronium and formoterol (BGF) metered dose inhaler (MDI) formulated with 3 different propellants: Propellant 1 (Treatment A [test]), Propellant 2 (Treatment B [test]) and Hydrofluoroalkane (HFA) (Treatment C [reference]).

DETAILED DESCRIPTION:
The study will comprise:

* Screening period: up to 28 days prior to first dosing;
* Three treatment periods of maximum 3 days each: participants will be resident from the morning of the day before the first dosing with BGF MDI (Day -1) in Treatment Period 1, throughout all treatment and washout periods up to discharge on Day 2 of Treatment Period 3;
* Follow-up: within 3 to 7 days after the last administration of BGF MDI. There will be a washout period of 3 to 7 days between each dose.

Each participant will receive 3 single-dose treatments of BGF MDI (1 dose Propellant 1 [Treatment A]; 1 dose Propellant 2 [Treatment B] and 1 dose HFA [Treatment C]), following an overnight fast of at least 8 hours. Each participant will be involved in the study for up to 53 days.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Non-smoking male participants with suitable veins for cannulation or repeated venipuncture.
* Participants must agree to follow the reproductive restrictions.
* Have a body mass index between 18 and 30 kg/m^2 and weigh at least 50 kg and no more than 100 kg.
* Participants must have a forced expiratory volume in one second ≥ 80% of the predicted value regarding age, height, and ethnicity at the screening visit.

Exclusion Criteria:

* History or current evidence of a clinically significant (CS) disease or disorder (including but not limited to cardiovascular, hepatic, renal, hematological, neurological, endocrine, gastrointestinal, or pulmonary).
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any CS illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational medicinal product (IMP).
* Narrow angle glaucoma not adequately treated. All medications approved for control of intraocular pressures are allowed, including topical ophthalmic non-selective β-blockers.
* Symptomatic prostatic hypertrophy or bladder neck obstruction/urinary retention that, in the opinion of the principal investigator (PI), is CS.
* Any cancer except squamous cell and basal cell carcinomas of the skin are allowed in the study.
* Any CS abnormalities in clinical chemistry, hematology, or urinalysis results, at screening and/or admission to the Clinical Unit:

  1. Systolic blood pressure (BP) < 90 mmHg or > 140 mmHg.
  2. Diastolic BP < 50 mmHg or > 90 mmHg.
  3. Heart rate < 45 or > 85 bpm.
* Any CS abnormal findings in vital signs, after 5 minutes supine rest, at screening and/or Day -1 of each Treatment Period, as judged by the PI.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting electrocardiogram (ECG) and any clinically important abnormalities in the 12-lead ECG as considered by the PI.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus antibody.
* Known or suspected history of drug abuse.
* Participant has a positive reverse transcription polymerase chain reaction test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) prior to randomization.
* Participant has clinical signs and symptoms consistent with SARS-CoV-2 infection (e.g., fever, dry cough, dyspnea, sore throat, fatigue, or laboratory confirmed acute infection with SARS-CoV-2).
* Participant who had severe course of coronavirus disease 2019 (COVID-19).
* Recent (within 14 days prior to admission to the Clinical Unit) exposure to someone who has COVID-19 symptoms or tested positive for SARS-CoV-2.
* Recent (within 14 days prior to admission to the Clinical Unit) visit to a healthcare facility where COVID-19 patients are being treated.
* Has a current occupation that involves routine exposure to potential COVID-19 patients or sources of SARS-CoV-2 infection.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study.
* Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to BGF.
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months prior to screening.
* Positive screen for drugs of abuse or cotinine at screening or on admission to the Clinical Unit or positive screen for alcohol at screening or on admission to the Clinical Unit.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
* Use of any prescribed or non-prescribed medication including antacids, analgesics, herbal remedies, megadose vitamins and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life.
* Known or suspected history of alcohol abuse or excessive intake of alcohol.
* Participants who have previously received BGF.
* Judgment by the PI that the participant should not participate in the study if they have any ongoing or recent minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Vulnerable participants, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
* History of any respiratory disorders such as asthma, COPD or idiopathic pulmonary fibrosis.
* Participants who cannot use an inhaler appropriately.
* Participants who cannot communicate reliably with the PI.
* Receipt of COVID-19 vaccine (regardless of vaccine delivery platform, eg vector, lipid nanoparticle) less than 7 days prior to the date of randomization (from last vaccination or booster dose).

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 47 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Han, Dr., Principal Investigator — PAREXEL Early Phase Clinical Unit-Los Angeles
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Aurivillius M, Bednarczyk A, Kokot M, Madriaga J, Mei J, Collison K, Surujbally R, Archbell J, Joshi V, Gillen M. Relative bioavailability of budesonide/glycopyrrolate/formoterol fumarate triple therapy delivered using next generation propellants with low global warming potential. Pulm Pharmacol Ther. 2023 Dec;83:102245. doi: 10.1016/j.pupt.2023.102245. Epub 2023 Aug 20. PMID 37607661
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5985C00001&attachmentIdentifier=7ae437a9-62d2-4284-bb3d-06a0a615cfeb&fileName=AZ_D5985C00001_(PXL_245780)_CSP.pdf&versionIdentifier=
- See also: CSP & SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5985C00001&attachmentIdentifier=00cd56e1-4a3c-40f6-93be-f56a6cbd0f64&fileName=AZ_D5985C00001_(PXL_245780)_Final_Protocol_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between 19 Oct 2020 to 17 May 2021 at a single study center - Parexel Early Phase Clinical Unit (Los Angeles).
Pre-assignment Details: This study consisted of a Screening Period of 28 days. There were three treatment periods of maximum three days each, with washout period of 3 to 7 days between each study dose administration. The assessments were done as per the schedule of assessment in the clinical study protocol.
Groups:
- Treatment Sequence ABC: Randomized participants received 3 single-dose treatments of budesonide, glycopyronnium, formoterol (BGF) metered dose inhaler (MDI) (1 dose Propellant 1 [Treatment A]; 1 dose Propellant 2 [Treatment B] and 1 dose HFA propellant [Treatment C]) in 3 treatment periods, with wash-out periods of 3 - 7 days between each study dose administration under fasted conditions.
- Treatment Sequence BCA: Randomized participants received 3 single-dose treatments of BGF MDI (1 dose Propellant 2 [Treatment B]; 1 dose HFA propellant [Treatment C] and 1 dose Propellant 1 [Treatment A]) in 3 treatment periods, with wash-out periods of 3 - 7 days between each study dose administration under fasted conditions.
- Treatment Sequence CAB: Randomized participants received 3 single-dose treatments of BGF MDI (1 dose HFA propellant [Treatment C]; 1 dose Propellant 1 [Treatment A] and 1 dose Propellant 2 [Treatment B]) in 3 treatment periods, with wash-out periods of 3 - 7 days between each study dose administration under fasted conditions.
- Treatment Sequence ACB: Randomized participants received 3 single-dose treatments of BGF MDI (1 dose Propellant 1 [Treatment A]; 1 dose HFA propellant [Treatment C] and 1 dose Propellant 2 [Treatment B]) in 3 treatment periods, with wash-out periods of 3 - 7 days between each study dose administration under fasted conditions.
- Treatment Sequence BAC: Randomized participants received 3 single-dose treatments of BGF MDI (1 dose Propellant 2 [Treatment B]; 1 dose Propellant 1 [Treatment A] and 1 dose HFA propellant [Treatment C]) in 3 treatment periods, with wash-out periods of 3 - 7 days between each study dose administration under fasted conditions.
- Treatment Sequence CBA: Randomized participants received 3 single-dose treatments of BGF MDI (1 dose HFA propellant [Treatment C]; 1 dose Propellant 2 [Treatment B] and 1 dose Propellant 1 [Treatment A]) in 3 treatment periods, with wash-out periods of 3 - 7 days between each study dose administration under fasted conditions.
Period: Overall Study
Arm/Group | Treatment Sequence ABC | Treatment Sequence BCA | Treatment Sequence CAB | Treatment Sequence ACB | Treatment Sequence BAC | Treatment Sequence CBA
Started | 8 | 8 | 8 | 8 | 7 | 8
Completed | 8 | 8 | 8 | 8 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Randomized Set consisted of all participants randomized into the study.
Groups:
- Treatment Sequence ABC: Randomized participants received 3 single-dose treatments of BGF MDI (1 dose Propellant 1 [Treatment A]; 1 dose Propellant 2 [Treatment B] and 1 dose HFA propellant [Treatment C]) in 3 treatment periods, with wash-out periods of 3 - 7 days between each study dose administration under fasted conditions.
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence ABC | Treatment Sequence BCA | Treatment Sequence CAB | Treatment Sequence ACB | Treatment Sequence BAC | Treatment Sequence CBA | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 8 | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.0 (7.56) | 38.5 (7.67) | 36.6 (6.63) | 34.4 (8.33) | 34.7 (11.63) | 39.1 (11.89) | 36.6 (8.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 8 | 8 | 8 | 8 | 7 | 8 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 1 | 1 | 2 | 2 | 11
  Not Hispanic or Latino | 5 | 6 | 7 | 7 | 5 | 6 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Black or African American | 2 | 3 | 3 | 4 | 3 | 3 | 18
  White | 6 | 3 | 5 | 2 | 3 | 3 | 22
  Other | 0 | 2 | 0 | 1 | 0 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of BGF MDI
Description: Evaluation of the relative bioavailability between the test formulations and the reference formulation for fixed dose combinations (FDCs) of BGF when delivered as BGF MDI with 3 different propellants by Cmax.
Time Frame: Pre-dose and 2, 5, 10, 20, 30, and 45 minutes post-dose and 1, 2, 4, 8, 12 and 24 hours post-dose
Population: The PK Analysis Set consisted of all participants in the Safety Analysis Set for whom at least 1 of the primary PK parameters could have been calculated, and who had no important protocol deviations thought to impact on the analysis of the PK data. Number Analyzed in each row signifies only the participants with available data that were analyzed for BGF MDI.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Groups:
- Treatment A: Participants received 2 inhalations of BGF MDI with Propellant 1 - test formulation (Treatment A)
- Treatment B: Participants received 2 inhalations of BGF MDI with Propellant 2 - test formulation (Treatment B)
- Treatment C: Participants received 2 inhalations of BGF MDI with HFA Propellant - reference formulation (Treatment C)
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 22 | 23
pg/mL
  Budesonide | 552.2 (54.74) | 483.2 (48.43) | 489.4 (61.61)
  Glycopyrronium | 11.74 (72.16) | 10.19 (58.42) | 10.76 (70.78)
  Formoterol | 12.70 (50.52) | 11.68 (47.22) | 11.48 (52.95)
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Statistical Comparison of Budesonide PK Parameters for Treatment A (test) versus Treatment C (reference); Test type: Other — Results based on linear mixed-effects analysis of variance model; Geometric mean Ratio (%) = 111.7, 90% CI 2-sided [91.01 to 137.1]
Statistical Analysis 2: Comparison: Treatment B vs Treatment C; Statistical Comparison of Budesonide PK Parameters for Treatment B (test) versus Treatment C (reference); Test type: Other — Results based on linear mixed-effects analysis of variance model; Geometric mean Ratio (%) = 98.78, 90% CI 2-sided [78.67 to 124.0]
Statistical Analysis 3: Comparison: Treatment A vs Treatment C; Statistical Comparison of Glycopyrronium PK Parameters for Treatment A (test) versus Treatment C (reference); Test type: Other — Results based on linear mixed-effects analysis of variance model; Geometric mean Ratio (%) = 108.3, 90% CI 2-sided [85.50 to 137.3]
Statistical Analysis 4: Comparison: Treatment B vs Treatment C; Statistical Comparison of Glycopyrronium PK Parameters for Treatment B (test) versus Treatment C (reference); Test type: Other — Results based on linear mixed-effects analysis of variance model; Geometric mean Ratio (%) = 94.88, 90% CI 2-sided [74.69 to 120.5]
Statistical Analysis 5: Comparison: Treatment A vs Treatment C; Statistical Comparison of Formoterol PK Parameters for Treatment A (test) versus Treatment C (reference); Test type: Other — Results based on linear mixed-effects analysis of variance model; Geometric mean Ratio (%) = 109.1, 90% CI 2-sided [97.02 to 122.7]
Statistical Analysis 6: Comparison: Treatment B vs Treatment C; Statistical Comparison of Formoterol PK Parameters for Treatment B (test) versus Treatment C (reference); Test type: Other — Results based on linear mixed-effects analysis of variance model; Geometric mean Ratio (%) = 100.1, 90% CI [83.78 to 119.5]

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinity (AUCinf) of BGF MDI
Description: Evaluation of the relative bioavailability between the test formulations and the reference formulation for FDCs of BGF when delivered as BGF MDI with 3 different propellants by AUCinf.
Time Frame: Pre-dose and 2, 5, 10, 20, 30, and 45 minutes post-dose and 1, 2, 4, 8, 12 and 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 22 | 21
h*pg/mL
  Budesonide | 2454 (36.76) | 2262 (32.27) | 2314 (45.60)
  Glycopyrronium: number analyzed (Participants) | 4 | 3 | 2
  Glycopyrronium | 30.32 (39.74) | 27.23 (30.67) | NA (NA) — Three values were required as a minimum for PK parameters to be summarized as per protocol.
  Formoterol: number analyzed (Participants) | 10 | 6 | 13
  Formoterol | 93.68 (35.71) | 115.1 (30.99) | 92.84 (30.45)
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Statistical Comparison of Budesonide PK Parameters for Treatment A (test) versus Treatment C (reference); Test type: Other — Results based on linear mixed-effects analysis of variance model; Geometric mean Ratio (%) = 104.7, 90% CI 2-sided [91.95 to 119.2]
Statistical Analysis 2: Comparison: Treatment B vs Treatment C; Statistical Comparison of Budesonide PK Parameters for Treatment B (test) versus Treatment C (reference); Test type: Other — Results based on linear mixed-effects analysis of variance model; Geometric mean Ratio (%) = 98.03, 90% CI 2-sided [83.33 to 115.3]
Statistical Analysis 3: Comparison: Treatment A vs Treatment C; Statistical Comparison of Formoterol PK Parameters for Treatment A (test) versus Treatment C (reference); Test type: Other — Results based on linear mixed-effects analysis of variance model; Geometric mean Ratio (%) = 96.00, 90% CI [70.33 to 131.0]
Statistical Analysis 4: Comparison: Treatment B vs Treatment C; Statistical Comparison of Formoterol PK Parameters for Treatment B (test) versus Treatment C (reference); Test type: Other — Results based on linear mixed-effects analysis of variance model; Geometric mean Ratio (%) = 116.7, 90% CI [86.31 to 157.8]

3. Primary Outcome: Area Under the Plasma Concentration- Curve From Time Zero to the Time of Last Quantifiable Concentration (AUClast) of BGF MDI
Description: Evaluation of the relative bioavailability between the test formulations and the reference formulation for FDCs of BGF when delivered as BGF MDI with 3 different propellants by AUClast.
Time Frame: Pre-dose and 2, 5, 10, 20, 30, and 45 minutes post-dose and 1, 2, 4, 8, 12 and 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 22 | 23
h*pg/mL
  Budesonide | 2391 (36.77) | 2197 (32.81) | 2232 (44.14)
  Glycopyrronium | 29.87 (88.09) | 28.63 (53.90) | 29.20 (82.24)
  Formoterol | 66.17 (50.54) | 74.34 (41.35) | 67.82 (55.58)
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Statistical Comparison of Budesonide PK Parameters for Treatment A (test) versus Treatment C (reference); Test type: Other — Results based on linear mixed-effects analysis of variance model; Geometric mean Ratio (%) = 107.3, 90% CI 2-sided [94.53 to 121.9]
Statistical Analysis 2: Comparison: Treatment B vs Treatment C; Statistical Comparison of Budesonide PK Parameters for Treatment B (test) versus Treatment C (reference); Test type: Other — Results based on linear mixed-effects analysis of variance model; Geometric mean Ratio (%) = 98.80, 90% CI 2-sided [84.59 to 115.4]
Statistical Analysis 3: Comparison: Treatment A vs Treatment C; Statistical Comparison of Glycopyrronium PK Parameters for Treatment A (test) versus Treatment C (reference); Test type: Other — Results based on linear mixed-effects analysis of variance model; Geometric mean Ratio (%) = 106.1, 90% CI 2-sided [86.18 to 130.6]
Statistical Analysis 4: Comparison: Treatment B vs Treatment C; Statistical Comparison of Glycopyrronium PK Parameters for Treatment B (test) versus Treatment C (reference); Test type: Other — Results based on linear mixed-effects analysis of variance model; Geometric mean Ratio (%) = 99.71, 90% CI 2-sided [80.84 to 123.0]
Statistical Analysis 5: Comparison: Treatment A vs Treatment C; Statistical Comparison of Formoterol PK Parameters for Treatment A (test) versus Treatment C (reference); Test type: Other — Results based on linear mixed-effects analysis of variance model; Geometric mean Ratio (%) = 98.13, 90% CI 2-sided [86.44 to 111.4]
Statistical Analysis 6: Comparison: Treatment B vs Treatment C; Statistical Comparison of Formoterol PK Parameters for Treatment B (test) versus Treatment C (reference); Test type: Other — Results based on linear mixed-effects analysis of variance model; Geometric mean Ratio (%) = 107.0, 90% CI 2-sided [88.82 to 128.9]

4. Secondary Outcome: Time to Reach Maximum Observed Concentration (Tmax) of BGF MDI
Description: Assessment of tmax of BGF when administered as 3 different propellant formulations.
Time Frame: Pre-dose and 2, 5, 10, 20, 30, and 45 minutes post-dose and 1, 2, 4, 8, 12 and 24 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 22 | 23
hours
  Budesonide | 0.50 [0.08 to 2.00] | 0.75 [0.08 to 2.00] | 0.52 [0.08 to 1.02]
  Glycopyrronium | 0.08 [0.03 to 0.75] | 0.08 [0.03 to 2.00] | 0.08 [0.03 to 2.00]
  Formoterol | 0.17 [0.08 to 2.00] | 0.50 [0.08 to 2.00] | 0.17 [0.07 to 2.00]

5. Secondary Outcome: Terminal Elimination Half-life (t½λz) of BGF MDI
Description: Assessment of t½λz of BGF when administered as 3 different propellant formulations.
Time Frame: Pre-dose and 2, 5, 10, 20, 30, and 45 minutes post-dose and 1, 2, 4, 8, 12 and 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 17 | 15 | 15
hours
  Budesonide | 4.420 (0.4003) | 4.438 (0.7886) | 4.574 (0.4267)
  Glycopyrronium: number analyzed (Participants) | 0 | 0 | 0
  Formoterol: number analyzed (Participants) | 1 | 0 | 1
  Formoterol | NA (NA) — Three values were required as a minimum for PK parameters to be summarized as per protocol. |  | NA (NA) — Three values were required as a minimum for PK parameters to be summarized as per protocol.

6. Secondary Outcome: Apparent Total Body Clearance of Drug After Extravascular Administration (CL/F) of BGF MDI
Description: Assessment of CL/F of BGF when administered as 3 different propellant formulations.
Time Frame: Pre-dose and 2, 5, 10, 20, 30, and 45 minutes post-dose and 1, 2, 4, 8, 12 and 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Litre/hour
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 22 | 21
Litre/hour
  Budesonide | 137.9 (43.28) | 148.6 (50.91) | 155.3 (105.4)
  Glycopyrronium: number analyzed (Participants) | 4 | 3 | 2
  Glycopyrronium | 502.6 (201.8) | 544.5 (158.1) | NA (NA) — Three values were required as a minimum for PK parameters to be summarized as per protocol.
  Formoterol: number analyzed (Participants) | 10 | 6 | 13
  Formoterol | 108.8 (43.64) | 87.14 (32.16) | 108.3 (38.41)

7. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase After Extravascular Administration (Vz/F) of BGF MDI
Description: Assessment of Vz/F of BGF when administered as 3 different propellant formulations.
Time Frame: Pre-dose and 2, 5, 10, 20, 30, and 45 minutes post-dose and 1, 2, 4, 8, 12 and 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 22 | 21
Litre
  Budesonide | 941.9 (328.6) | 1023 (330.4) | 1142 (1005)
  Glycopyrronium: number analyzed (Participants) | 4 | 3 | 2
  Glycopyrronium | 1992 (200.5) | 2079 (638.9) | NA (NA) — Three values were required as a minimum for PK parameters to be summarized as per protocol.
  Formoterol: number analyzed (Participants) | 10 | 6 | 13
  Formoterol | 1171 (281.2) | 1007 (211.3) | 1167 (180.9)

8. Secondary Outcome: Number of Participants With Serious Adverse Events (SAE) and Non-serious Adverse Events
Description: Assessment of the safety and tolerability of a combination of BGF when administered as single doses in 3 different propellant formulations in healthy participants.
Time Frame: Screening, Day -1 until Follow-up visit, up to 53 days
Population: The Safety Analysis Set included all participants who received at least 1 inhalation of any BGF MDI formulated treatment. This included all original and replacement participants where the 1 inhalation criterion was met.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 47 | 47 | 47
Participants
  Any AE | 9 | 10 | 10
  Any AE with outcome = death | 0 | 0 | 0
  Any serious AE (including events with outcome = death) | 0 | 0 | 0
  Any AE leading to discontinuation of IMP | 0 | 0 | 0
  Any AE leading to withdrawal from study | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening, Day -1 until Follow-up visit, up to 53 days
Arm/Group | Treatment A | Treatment B | Treatment C
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 9/47 | 10/47 | 10/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=47) | Treatment B (N=47) | Treatment C (N=47)
Headache (Nervous system disorders) | 2 | 2 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Medical device site dermatitis (General disorders) | 1 | 1 | 2
Chest discomfort (General disorders) | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 0 | 1
Hypermetropia (Eye disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information may be disclosed without prior written approval from AstraZeneca AB.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT04600505/Prot_SAP_000.pdf